CLINICAL TRIAL: NCT04314232
Title: Changes in Organ Specific Biomarkers, Virus Expression and Prognosis of Covid-19
Brief Title: Mechanisms for Covid-19 Disease Complications
Acronym: COVID MECH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor, University Hospital, Akershus
Other Study IDs: 117589
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: COVID; Coronavirus Infection
Keywords: Covid-19; Biomarkers; Cardiovascular disease; Prognosis
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 is associated with a wide range of symptoms and clinical trajectories, and early identification of patients at risk for developing severe disease is desirable. Several risk markers and comorbidity profiles have been proposed but their relative importance in unselected patients admitted to hospital with Covid-19 remains unclear. This study aims to assess the prognostic value organ specific biomarkers, viral dynamics and immune response markers in patients infected with SARS-CoV2.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years of age with a positive test for SARS-CoV2 are eligble for inclusion.
* Healty age-matched volunteers will be included as a control group

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with a positive test for SARS-CoV2 admitted to Akershus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ICU admission or death | From hospital admission (baseline) until the date of either admission to the ICU or death during the index hospitalization (up to 52 weeks)
  Combined outcome measure of either ICU admission or death

SECONDARY OUTCOMES:
Number of participants with ICU admission | From hospital admission (baseline) until the date of admission to the ICU during the index hospitalization (up to 52 weeks)
  ICU admission
Number of participants with death from all causes | From hospital admission (baseline) unitl the date of death during the index hospitalization (up to 52 weeks)
  Hospital mortality
Total duration of ICU stay | From admission to the ICU until transfer to another ward, discharge from the hospital or death during the index hospitalization (up to 52 weeks)
  Total time admitted to the ICU
Total duration of hospital stay | From hospital admission (baseline) until hospital discharge or death during the index hospitalization (up to 52 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Derived] Omland T, Prebensen C, Jonassen C, Svensson M, Berdal JE, Seljeflot I, Myhre PL. Soluble ST2 concentrations associate with in-hospital mortality and need for mechanical ventilation in unselected patients with COVID-19. Open Heart. 2021 Dec;8(2):e001884. doi: 10.1136/openhrt-2021-001884. PMID 34933965
- [Derived] Myhre PL, Heck SL, Skranes JB, Prebensen C, Jonassen CM, Berge T, Mecinaj A, Melles W, Einvik G, Ingul CB, Tveit A, Berdal JE, Rosjo H, Lyngbakken MN, Omland T. Cardiac pathology 6 months after hospitalization for COVID-19 and association with the acute disease severity. Am Heart J. 2021 Dec;242:61-70. doi: 10.1016/j.ahj.2021.08.001. Epub 2021 Aug 13. PMID 34400140
- [Derived] Myhre PL, Prebensen C, Jonassen CM, Berdal JE, Omland T. SARS-CoV-2 Viremia is Associated With Inflammatory, But Not Cardiovascular Biomarkers, in Patients Hospitalized for COVID-19. J Am Heart Assoc. 2021 May 4;10(9):e019756. doi: 10.1161/JAHA.120.019756. Epub 2021 Feb 18. PMID 33596668
- [Derived] Myhre PL, Prebensen C, Strand H, Roysland R, Jonassen CM, Rangberg A, Sorensen V, Sovik S, Rosjo H, Svensson M, Berdal JE, Omland T. Growth Differentiation Factor 15 Provides Prognostic Information Superior to Established Cardiovascular and Inflammatory Biomarkers in Unselected Patients Hospitalized With COVID-19. Circulation. 2020 Dec;142(22):2128-2137. doi: 10.1161/CIRCULATIONAHA.120.050360. Epub 2020 Oct 15. PMID 33058695